CLINICAL TRIAL: NCT03036488
Title: A Phase III, Randomized, Double-blind Study to Evaluate Pembrolizumab Plus Chemotherapy vs Placebo Plus Chemotherapy as Neoadjuvant Therapy and Pembrolizumab vs Placebo as Adjuvant Therapy for Triple Negative Breast Cancer (TNBC)
Brief Title: Study of Pembrolizumab (MK-3475) Plus Chemotherapy vs Placebo Plus Chemotherapy as Neoadjuvant Therapy and Pembrolizumab vs Placebo as Adjuvant Therapy in Participants With Triple Negative Breast Cancer (TNBC) (MK-3475-522/KEYNOTE-522)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-522; 173567 (Registry Identifier: JAPIC-CTI); MK-3475-522 (Other: MSD); KEYNOTE-522 (Other: MSD); 2022-501382-49-00 (Registry Identifier: EU CT); U1111-1280-2361 (Registry Identifier: UTN); 2016-004740-11 (EudraCT Number)
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — pembrolizumab; Carboplatin; Paclitaxel; Doxorubicin; Epirubicin; Cyclophosphamide; Filgrastim; pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Chemotherapy (Experimental): Participants receive pembrolizumab every 3 weeks (Q3W) + paclitaxel weekly + carboplatin (weekly or Q3W) x 4 cycles, followed by pembrolizumab Q3W + (doxorubicin OR epirubicin) + cyclophosphamide Q3W x 4 cycles as neoadjuvant therapy prior to surgery; followed by 9 cycles of pembrolizumab Q3W as adjuvant therapy post-surgery. Each cycle is 21 days.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Epirubicin; Drug: Cyclophosphamide; Biological: Granulocyte colony stimulating factor: Filgrastim or Pegfilgastrim
- Placebo + Chemotherapy (Active Comparator): Participants receive placebo (normal saline solution) Q3W + paclitaxel weekly + carboplatin (weekly or Q3W) x 4 cycles, followed by placebo + (doxorubicin OR epirubicin) + cyclophosphamide Q3W x 4 cycles as neoadjuvant therapy prior to surgery; followed by 9 cycles of placebo Q3W as adjuvant therapy post-surgery. Each cycle is 21 days.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Placebo; Biological: Granulocyte colony stimulating factor: Filgrastim or Pegfilgastrim

INTERVENTIONS:
Biological: Pembrolizumab — On Day 1 of each cycle in the neoadjuvant and adjuvant phases of the study for a total of 17 cycles; intravenous (IV) infusion.
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab + Chemotherapy
Drug: Carboplatin — On Day 1 of Cycles 1-4 of the neoadjuvant phase of the study OR on Days 1, 8, 15 of Cycles 1-4 of the neoadjuvant phase of the study; IV infusion.
  Other Names: PARAPLATIN®
Drug: Paclitaxel — On Days 1, 8 and 15 of Cycles 1-4 in the neoadjuvant phase of the study; IV infusion.
  Other Names: TAXOL®
Drug: Doxorubicin — On Day 1 of Cycles 5-8 of the neoadjuvant phase of the study; IV injection.
  Other Names: ADRIAMYCIN®
Drug: Epirubicin — On Day 1 of Cycles 5-8 of the neoadjuvant phase of the study; IV injection.
  Other Names: ELLENCE®
Drug: Cyclophosphamide — On Day 1 of Cycles 5-8 of the neoadjuvant phase of the study; IV infusion.
  Other Names: CYTOXAN®
Drug: Placebo — normal saline solution or dextrose: On Day 1 of each cycle in the neoadjuvant and adjuvant phases of the study for a total of 17 cycles; IV infusion
  Arms: Placebo + Chemotherapy
Biological: Granulocyte colony stimulating factor: Filgrastim or Pegfilgastrim — For prevention of neutropenia, filgrastim 5 μg/kg/day via subcutaneous (SC) injection administered per standard of care after chemotherapy OR pegfilgastrim 100 µg/kg (individualized) or 6 mg (general approach) via SC injection administered per standard of care.
  Other Names: NEUPOGEN®; NEULASTA®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pembrolizumab (MK-3475) plus chemotherapy vs placebo plus chemotherapy as neoadjuvant therapy and pembrolizumab vs placebo as adjuvant therapy in participants who have triple negative breast cancer (TNBC).

After a screening phase of approximately 28 days, each participant will receive neoadjuvant study treatment (Pembrolizumab + Chemotherapy OR Placebo + Chemotherapy) based on the randomization schedule for approximately 24 weeks (8 cycles). Each participant will then undergo definitive surgery 3-6 weeks after conclusion of the last cycle of the neoadjuvant study treatment. After definitive surgery, each participant will receive adjuvant study treatment (Pembrolizumab OR Placebo) for approximately 27 weeks (9 cycles). Following adjuvant study treatment, each participant will be monitored for safety, survival and disease recurrence.

The primary study hypothesis is that pembrolizumab is superior to placebo, in combination with chemotherapy, as measured by the rate of Pathological Complete Response (pCR) and/or Event-free Survival (EFS), in participants with locally advanced TNBC.

ELIGIBILITY:
Inclusion Criteria:

* Has newly diagnosed, locally advanced, centrally confirmed TNBC, as defined by the most recent American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines.
* Has previously untreated locally advanced non-metastatic (M0) TNBC defined as the following combined primary tumor (T) and regional lymph node (N) staging per current American Joint Committee of Cancer (AJCC) staging criteria for breast cancer as assessed by the investigator based on radiological and/or clinical assessment:

  * T1c, N1-N2
  * T2, N0-N2
  * T3, N0-N2
  * T4a-d, N0-N2
* Provides a core needle biopsy consisting of at least 2 separate tumor cores from the primary tumor at screening to the central laboratory.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 performed within 10 days of treatment initiation.
* Demonstrates adequate organ function.
* Males and female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 12 months after the last dose of study treatment for participants who have received cyclophosphamide, and 6 months after the last dose of study treatment for participants who did not.

Exclusion Criteria:

* Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Has received prior chemotherapy, targeted therapy, and radiation therapy within the past 12 months.
* Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death - ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated antigen-4 [CTLA-4], OX-40, CD137 [tumor necrosis factor receptor superfamily member 9 (TNFRSF9)]) or has previously participated in a pembrolizumab (MK-3475) clinical study.
* Is currently participating in or has participated in an interventional clinical study with an investigational compound or device within 4 weeks of the first dose of treatment in this current study.
* Has received a live vaccine within 30 days of the first dose of study treatment.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (i.e., dosing exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or Hepatitis C.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has significant cardiovascular disease, such as: history of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last 6 months OR congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV or history of CHF NYHA Class III or IV.
* Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study, starting with the screening visit through 12 months after the last dose of study treatment for participants who have received cyclophosphamide, and for 6 months after the last dose of study treatment for participants who have not.
* Has a known hypersensitivity to the components of the study treatment or its analogs.
* Has a known history of active tuberculosis (TB, Bacillus Tuberculosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1174 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | Up to approximately 27-30 weeks
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current American Joint Committee on Cancer (AJCC) staging criteria assessed by the local pathologist at the time of definitive surgery.
Event-free Survival (EFS) as assessed by Investigator | Up to approximately 8 years
  EFS is defined as the time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.

SECONDARY OUTCOMES:
pCR rate using an alternative definition, ypT0 ypN0 (i.e., no invasive or noninvasive residual in breast or nodes) at the time of definitive surgery | Up to approximately 27-30 weeks
  pCR rate (ypT0 ypN0) is defined as the percentage of participants without residual invasive and in situ cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants and in participants with tumors expressing Programmed Death-Ligand 1 (PD-L1).
pCR rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | Up to approximately 27-30 weeks
  pCR rate (ypT0/Tis) is defined as the percentage of participants without invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in participants with tumors expressing PD-L1.
EFS in participants with tumors expressing PD-L1 | Up to approximately 8 years
  EFS is defined as the time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
pCR rate using an alternative definition, ypT0/Tis (i.e., absence of invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement) at the time of definitive surgery | Up to approximately 27-30 weeks
  pCR rate (ypT0/Tis) is defined as the percentage of participants without invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants and in participants with tumors expressing PD-L1.
Overall survival (OS) | Up to approximately 8 years
  OS is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis will be censored at the date of the last follow-up.
Percentage of participants who experience an adverse event (AE) | Up to approximately 61 weeks
  An AE is defined as any untoward medical occurrence in a participant administered study treatment which does not necessarily have to have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment or protocol-specified procedure, whether or not considered related to study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE.
Percentage of participants who discontinue study treatment due to an AE | Up to approximately 57 weeks
  An AE is defined as any untoward medical occurrence in a participant administered study treatment which does not necessarily have to have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment or protocol-specified procedure, whether or not considered related to study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE.
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Core 30 Questionnaire (QLQ-C30) score | Up to approximately 27-30 weeks
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Individual responses are given on a 4-point scale (1=Not at All to 4=Very Much), with a lower score indicating a better outcome. The EORTC-QLQ-C30 score will be presented for all participants and for participants with tumors expressing PD-L1.
EORTC Breast Cancer-Specific QoL Questionnaire (QLQ-BR23) score | Up to approximately 27-30 weeks
  The EORTC-QLQ-BR23 is a 23-item questionnaire developed to assess the quality of life of breast cancer patients. Individual responses are given on a 4-point scale (1=Not at All to 4=Very Much), with a lower score indicating a better outcome. The EORTC-QLQ-BR23 score will be presented for all participants and for participants with tumors expressing PD-L1.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (193):
- United States (47):
  - Virginia G. Piper Cancer Center Pharmacy - Scottsdale Healthcare ( Site 0089), Scottsdale, Arizona
  - Arizona Oncology Associates PC- HOPE ( Site 8001), Tucson, Arizona
  - Cedars Sinai Medical Center ( Site 0091), Los Angeles, California
  - Pacific Cancer Care ( Site 0069), Monterey, California
  - ICRI ( Site 0072), Whittier, California
  - University of Colorado Cancer Center ( Site 0021), Aurora, Colorado
  - Yale University School of Medicine ( Site 0054), New Haven, Connecticut
  - Christiana Hospital ( Site 0029), Newark, Delaware
  - Univ of Miami-Sylvester Comprehensive Cancer Center- Kendall satellite ( Site 0079), Miami, Florida
  - The University of Chicago Medical Center ( Site 0047), Chicago, Illinois
  - North Shore University Health System ( Site 0081), Evanston, Illinois
  - Orchard Healthcare Research Inc. ( Site 0049), Skokie, Illinois
  - Goshen Center for Cancer Care ( Site 0010), Goshen, Indiana
  - University of Iowa Hospital and Clinics ( Site 0038), Iowa City, Iowa
  - New England Cancer Specialists ( Site 0005), Scarborough, Maine
  - Henry Ford Hospital ( Site 0003), Detroit, Michigan
  - Minnesota Oncology Hematology, PA ( Site 8013), Minneapolis, Minnesota
  - Rutgers Cancer Institute of New Jersey ( Site 0073), New Brunswick, New Jersey
  - Broome Oncology, LLC ( Site 8002), Johnson City, New York
  - Nyack Hospital Infusion Center ( Site 0059), Nyack, New York
  - TriHealth Cancer Institute-Good Samaritan Hospital ( Site 0044), Cincinnati, Ohio
  - Oncology Hematology Care, Inc. ( Site 8011), Cincinnati, Ohio
  - Providence Portland Medical Center ( Site 0052), Portland, Oregon
  - Northwest Cancer Specialists, P.C. ( Site 8008), Portland, Oregon
  - Magee - Women's Hospital ( Site 0011), Pittsburgh, Pennsylvania
  - Rhode Island Hospital ( Site 0060), Providence, Rhode Island
  - The West Clinic, P.C. ( Site 0078), Germantown, Tennessee
  - Texas Oncology-Austin Central ( Site 8005), Austin, Texas
  - Parkland Health and Hospital System ( Site 0093), Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center ( Site 8006), Dallas, Texas
  - Simmons Cancer Center ( Site 0094), Dallas, Texas
  - UT Southwestern Medical Center ( Site 0030), Dallas, Texas
  - Moncrief Cancer Institute ( Site 0092), Fort Worth, Texas
  - Texas Oncology-Memorial City ( Site 8003), Houston, Texas
  - Houston Methodist Cancer Center ( Site 0013), Houston, Texas
  - Texas Oncology- Plano East ( Site 8010), Plano, Texas
  - Texas Oncology-San Antonio Northeast ( Site 8012), San Antonio, Texas
  - Texas Oncology-Tyler ( Site 8007), Tyler, Texas
  - University of Virginia ( Site 0022), Charlottesville, Virginia
  - Virginia Cancer Specialists, PC ( Site 8009), Fairfax, Virginia
  - Bon Secours Cancer Institute Medical Oncology at St. Mary's ( Site 0033), Midlothian, Virginia
  - Peninsula Cancer Institute, LLC ( Site 0041), Newport News, Virginia
  - Virginia Oncology Associates ( Site 8000), Norfolk, Virginia
  - Kadlec Clinic Hematology and Oncology ( Site 0087), Kennewick, Washington
  - Seattle Cancer Care Alliance ( Site 0068), Seattle, Washington
  - Medical Oncology Associates (Summit Cancer Centers) ( Site 0014), Spokane, Washington
  - YVMH dba Vrigina Mason Memorial/North Star Lodge Cancer Center ( Site 8004), Yakima, Washington
- Australia (7):
  - Royal North Shore Hospital ( Site 2000), Sydney, New South Wales
  - Westmead Hospital ( Site 2002), Sydney, New South Wales
  - Royal Adelaide Hospital ( Site 2008), Adelaide, South Australia
  - Cabrini Health ( Site 2009), Malvern East, Victoria
  - Frankston Hospital ( Site 2010), Franskton
  - Royal Brisbane and Women s Hospital ( Site 2003), Herston
  - St John of God Subiaco Hospital ( Site 2006), Perth
- Brazil (9):
  - Hospital Nossa Senhora da Conceicao ( Site 0203), Porto Alegre, Rio Grande do Sul
  - UOPECCAN - Uniao Oeste Paranaense de Estudos e Combate ao Cancer ( Site 0206), Cascavel
  - Universidade de Caxias do Sul ( Site 0201), Caxias do Sul
  - Hospital Erasto Gaertner ( Site 0207), Curitiba
  - Instituto do Cancer do Ceara ( Site 0205), Fortaleza
  - Hospital Araujo Jorge ( Site 0204), Goiânia
  - Hospital Sao Lucas da PUCRS ( Site 0200), Porto Alegre
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto ( Site 0208), São José do Rio Preto
  - Instituto do Cancer de Sao Paulo - ICESP ( Site 0211), São Paulo
- Canada (7):
  - Tom Baker Cancer Centre ( Site 0105), Calgary, Alberta
  - The Ottawa Hospital - Cancer Care ( Site 0100), Ottawa, Ontario
  - Princess Margaret Cancer Centre ( Site 0103), Toronto, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0106), Montreal, Quebec
  - Jewish General Hospital ( Site 0101), Montreal, Quebec
  - CHU de Quebec Universite Laval - Hopital du Saint-Sacrement ( Site 0104), Québec, Quebec
  - CIUSSS de l'Estrie-CHUS ( Site 0102), Sherbrooke, Quebec
- Colombia (6):
  - Oncomedica S.A. ( Site 0404), Montería, Departamento de Córdoba
  - Oncologos del Occidente S.A. ( Site 0405), Pereira, Risaralda Department
  - Hospital Universitario San Ignacio ( Site 0401), Bogotá
  - Instituto Nacional de Cancerologia [Bogota-Colombia] ( Site 0403), Bogotá
  - Hemato Oncologos S.A. ( Site 0400), Cali
  - Instituto De Cancerologia S.A. ( Site 0406), Medellín
- France (11):
  - CHU Jean Minjoz ( Site 0917), Besançon
  - Polyclinique Bordeaux Nord Aquitaine ( Site 0911), Bordeaux
  - Centre Francois Baclesse ( Site 0907), Caen
  - Centre Jean Perrin ( Site 0903), Clermont-Ferrand
  - Clinique Victor Hugo ( Site 0901), Le Mans
  - Hopital prive du Confluent ( Site 0902), Nantes
  - Institut Curie ( Site 0909), Paris
  - Hopital Saint Louis ( Site 0908), Paris
  - Hopital Diaconesses Croix Saint Simon ( Site 0905), Paris
  - CHU de la Miletrie Poitiers ( Site 0913), Poitiers
  - Institut Claudius Regaud IUCT Oncopole ( Site 0914), Toulouse
- Germany (9):
  - HELIOS Klinikum Berlin-Buch ( Site 1005), Berlin
  - Gynaekologisches Zentrum ( Site 1004), Bonn
  - Universitaetsklinikum Erlangen ( Site 1001), Erlangen
  - Kliniken Essen Mitte ( Site 1012), Essen
  - Universitaetsklinik und Poliklinik Halle/Saale ( Site 1008), Halle
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 1007), Hamburg
  - Klinikum der Universit. Muenchen ( Site 1002), München
  - Caritasklinik St. Theresia ( Site 1011), Saarbrücken
  - Universitaets-Frauenklinik Tuebingen ( Site 1003), Tübingen
- Ireland (2):
  - Bon Secours Hospital ( Site 1551), Cork
  - St Vincents University Hospital ( Site 1550), Dublin
- Israel (6):
  - Assaf Harofeh MC ( Site 1605), Beer Yaakov-Zerifin
  - Oncology institute ( Site 1601), Beersheba
  - Hadassah Ein Karem - Sharett Institute of Oncology ( Site 1600), Jerusalem
  - Rabin-Medical Center ( Site 1604), Petah Tikva
  - Sheba Medical Center ( Site 1602), Ramat Gan
  - Sourasky Medical Center ( Site 1603), Tel Aviv
- Italy (6):
  - Istituto Scientifico Romagnolo per Studio e Cura Tumori IRST ( Site 1101), Meldola, FC
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia ( Site 1103), Brescia
  - Ospedale San Luca, AZIENDA USL2 TOSCANA NORD OVEST ( Site 1105), Lucca
  - Ospedale Civile di Macerata ( Site 1104), Macerata
  - Istituto Europeo di Oncologia ( Site 1106), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 1102), Napoli
- Japan (19):
  - Aichi Cancer Center Hospital ( Site 2502), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 2518), Kashiwa, Chiba
  - National Hospital Organization Hokkaido Cancer Center ( Site 2512), Sapporo, Hokkaido
  - Hyogo College of Medicine Hospital ( Site 2506), Nishinomiya, Hyōgo
  - Tokai University Hospital ( Site 2517), Isehara, Kanagawa
  - St. Marianna University School of Medicine Hospital ( Site 2516), Kawasaki, Kanagawa
  - Kindai University Hospital ( Site 2507), Sayama, Osaka
  - Saitama Medical University International Medical Center ( Site 2513), Hidaka, Saitama
  - Saitama Cancer Center ( Site 2510), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 2514), Sunto-gun, Shizuoka
  - Chiba Cancer Center ( Site 2519), Chiba
  - Hiroshima City Hiroshima Citizens Hospital ( Site 2501), Hiroshima
  - Social medical corporation Hakuaikai Sagara Hospital ( Site 2508), Kagoshima
  - Kumamoto University Hospital ( Site 2515), Kumamoto
  - National Hospital Organization Osaka National Hospital ( Site 2505), Osaka
  - National Cancer Center Hospital ( Site 2500), Tokyo
  - St.Luke's International Hospital ( Site 2511), Tokyo
  - Toranomon Hospital ( Site 2503), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 2509), Tokyo
- Poland (8):
  - Mazowiecki Szpital Onkologiczny ( Site 1713), Wieliszew, Masovian Voivodeship
  - Centrum Onkologii Instytut im. Marii Skłodowskiej Curie ( Site 1717), Gliwice, Silesian Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka ( Site 1708), Bydgoszcz
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka ( Site 1712), Bydgoszcz
  - Szpital Morski im. PCK. Szpitale Pomorskie Sp. Z o.o ( Site 1701), Gdynia
  - Centrum Onkologii Instytut im. Marii Sklodowskiej Curie ( Site 1719), Krakow
  - Centrum Onkologii Ziemi Lubelskiej im. sw. Jana z Dukli ( Site 1700), Lublin
  - Dolnoslaskie Centrum Onkologii. ( Site 1702), Wroclaw
- Portugal (3):
  - Fundacao Champalimaud ( Site 2444), Lisbon
  - Hospital de Santa Maria, E.P.E. ( Site 2445), Lisbon
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil E.P.E. ( Site 2446), Porto
- Russia (7):
  - Arkhangelsk Clinical Oncological Dispensary ( Site 1810), Arkhangelsk
  - Chelyabinsk Regional Clinical Oncological Dispensary ( Site 1805), Chelyabinsk
  - Republican Clinical Oncology Dispensary of Tatarstan MoH ( Site 1806), Kazan'
  - Russian Oncological Research Center n.a. N.N.Blokhin of MoH ( Site 1801), Moscow
  - GBU RO Regional Clinical Oncological Dispensary ( Site 1808), Ryazan
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 1803), Saint Petersburg
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan ( Site 1804), Ufa
- National Cancer Centre Singapore ( Site 2600), Singapore, Singapore
- South Korea (4):
  - Seoul National University Hospital ( Site 2101), Seoul
  - Severance Hospital Yonsei University Health System ( Site 2100), Seoul
  - Asan Medical Center ( Site 2102), Seoul
  - Samsung Medical Center ( Site 2103), Seoul
- Spain (10):
  - ICO L Hospitalet ( Site 1305), L'Hospitalet de Llobregat, Barcelona
  - Hospital Quiron de Madrid ( Site 1303), Pozuelo de Alarcón, Madrid
  - Hospital del Mar ( Site 1306), Barcelona
  - Instituto Oncologico Baselga.Hospital Quiron. ( Site 1312), Barcelona
  - Hospital General Universitari Vall d Hebron ( Site 1301), Barcelona
  - Hospital Universitario Reina Sofia ( Site 1304), Córdoba
  - Hospital Universitario Ramon y Cajal ( Site 1300), Madrid
  - Complejo Hospitalario Universitario de Santiago ( Site 1308), Santiago de Compostela
  - Hospital Universitario Virgen del Rocio ( Site 1314), Seville
  - Hospital Clinico Univ de Valencia ( Site 1313), Valencia
- Sweden (4):
  - Linkopings Universitetssjukhus ( Site 1402), Linköping
  - Karolinska Universitetssjukhuset Solna ( Site 1404), Solna
  - Norrlands Universitetssjukhus ( Site 1401), Umeå
  - Akademiska Sjukhuset ( Site 1403), Uppsala
- Taiwan (6):
  - Taipei Veterans General Hospital ( Site 2302), Taipei, Beitou
  - National Cheng Kung University Hospital ( Site 2305), Tainan
  - National Taiwan University Hospital ( Site 2301), Taipei
  - MacKay Memorial Hospital ( Site 2303), Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 2304), Taipei
  - Linkou Chang Gung Memorial Hospital ( Site 2300), Taoyuan District
- Turkey (Türkiye) (14):
  - Samsun Ondokuz Mayıs Universitesi Tıp Fakultesi Hastanesi ( Site 1910), Samsun, Atakum
  - Adana Acıbadem Hospital Department of Medical Oncology ( Site 1906), Adana
  - Baskent Unıversity Adana Kısla Hospital ( Site 1903), Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 1912), Ankara
  - Abdurrahman Yurtaslan Oncology Training and Research Hospital ( Site 1909), Ankara
  - Ozel Medicana International Ankara Hastanesi ( Site 1915), Ankara
  - Antalya Memorial Hospital Department of Medical Oncology ( Site 1908), Antalya
  - Trakya University Medical Faculty Balkan Oncology Hospital ( Site 1901), Edirne
  - İstanbul University Cerrahpaşa Medical Faculty ( Site 1904), Istanbul
  - Amerikan Hospital Medical ( Site 1902), Istanbul
  - Memorial Sisli Hastanesi ( Site 1913), Istanbul
  - Acibadem Altunizade Hastanesi ( Site 1900), Istanbul
  - Ege University Medical Faculty Tulay Aktas Oncology Hospital ( Site 1905), Izmir
  - Izmir Medical Park Hospital Department of Medical Oncology ( Site 1907), Izmir
- United Kingdom (7):
  - Colchester General Hospital ( Site 1508), Colchester, Essex
  - Barts Cancer Institute ( Site 1500), London
  - St George s Hospital ( Site 1516), London
  - Maidstone Hospital ( Site 1511), Maidstone
  - The James Cook University Hospital ( Site 1515), Middlesbrough
  - Nottingham University Hospitals NHS Trust ( Site 1505), Nottingham
  - Royal Cornwall Hospitals NHS Trust ( Site 1504), Truro

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Schmid P, Cortes J, Dent R, McArthur H, Pusztai L, Kummel S, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Im SA, Untch M, Fasching PA, Mouret-Reynier MA, Foukakis T, Ferreira M, Cardoso F, Zhou X, Karantza V, Tryfonidis K, Aktan G, O'Shaughnessy J; KEYNOTE-522 Investigators. Overall Survival with Pembrolizumab in Early-Stage Triple-Negative Breast Cancer. N Engl J Med. 2024 Nov 28;391(21):1981-1991. doi: 10.1056/NEJMoa2409932. Epub 2024 Sep 15. PMID 39282906
- [Derived] Takahashi M, Mukai H, Takano T, Tsugawa K, Inoue K, Itoh M, Watanabe J, Tanabe Y, Yamamoto N, Miyoshi Y, Watanabe K, Mukohara T, Kong Y, Shimura M, Beca F, Schmid P, Iwata H. Pembrolizumab for Early-Stage Triple-Negative Breast Cancer: KEYNOTE-522 Japan Subgroup Analysis. Cancer Sci. 2026 Jan 14. doi: 10.1111/cas.70307. Online ahead of print. PMID 41536071
- [Derived] Dent R, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Untch M, Fasching PA, Cardoso F, Haiderali A, Jia L, Nguyen AM, Pan W, O'Shaughnessy J, Schmid P. Neoadjuvant pembrolizumab plus chemotherapy/adjuvant pembrolizumab for early-stage triple-negative breast cancer: quality-of-life results from the randomized KEYNOTE-522 study. J Natl Cancer Inst. 2024 Oct 1;116(10):1654-1663. doi: 10.1093/jnci/djae129. PMID 38913881
- [Derived] Favre-Bulle A, Huang M, Haiderali A, Bhadhuri A. Cost-Effectiveness of Neoadjuvant Pembrolizumab plus Chemotherapy Followed by Adjuvant Pembrolizumab in Patients with High-Risk, Early-Stage, Triple-Negative Breast Cancer in Switzerland. Pharmacoecon Open. 2024 Jan;8(1):91-101. doi: 10.1007/s41669-023-00445-8. Epub 2023 Nov 24. PMID 37999854
- [Derived] Takahashi M, Cortes J, Dent R, Pusztai L, McArthur H, Kummel S, Denkert C, Park YH, Im SA, Ahn JH, Mukai H, Huang CS, Chen SC, Kim MH, Jia L, Li XT, Tryfonidis K, Karantza V, Iwata H, Schmid P. Pembrolizumab Plus Chemotherapy Followed by Pembrolizumab in Patients With Early Triple-Negative Breast Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2342107. doi: 10.1001/jamanetworkopen.2023.42107. PMID 37966841
- [Derived] Schmid P, Cortes J, Dent R, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Untch M, Fasching PA, Cardoso F, Andersen J, Patt D, Danso M, Ferreira M, Mouret-Reynier MA, Im SA, Ahn JH, Gion M, Baron-Hay S, Boileau JF, Ding Y, Tryfonidis K, Aktan G, Karantza V, O'Shaughnessy J; KEYNOTE-522 Investigators. Event-free Survival with Pembrolizumab in Early Triple-Negative Breast Cancer. N Engl J Med. 2022 Feb 10;386(6):556-567. doi: 10.1056/NEJMoa2112651. PMID 35139274
- [Derived] Perez-Garcia J, Soberino J, Racca F, Gion M, Stradella A, Cortes J. Atezolizumab in the treatment of metastatic triple-negative breast cancer. Expert Opin Biol Ther. 2020 Sep;20(9):981-989. doi: 10.1080/14712598.2020.1769063. Epub 2020 May 25. PMID 32450725
- [Derived] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26186&tenant=MT_MSD_9011